CLINICAL TRIAL: NCT01806454
Title: Calcium Supplementation to Prevent Preeclampsia in Sichuan Province of China: a Multi-center, Prospective Random Trial
Brief Title: Calcium Supplementation to Prevent Preeclampsia in Sichuan Province of China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Second University Hospital (Other)
Collaborators: Sichuan Academy of Medical Sciences (Other); Guang'an people's hospital of Sichuan province (Other); pengzhou shi fuyou baojianyuan (Unknown); The First People's Hospital of Neijiang (Other); Suining Central Hospital (Other); Sichuan Provincial Maternal and Child Health Care Hospital (Unknown); Chengdu Women's and Children's Central Hospital (Other)
Responsible Party: Principal Investigator, Xinghui Liu, Professor, West China Second University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: hx2ck1
Record Dates: First submitted 2013-03-01; First posted 2013-03-07 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2014-04

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Calcium

ARMS (2):
- calcium A (Active Comparator): tablets, 600mg per day,till birth
  Interventions: Drug: calcium
- calcium B (Active Comparator): tablets,1200mg per day,till birth
  Interventions: Drug: calcium

INTERVENTIONS:
Drug: calcium

SUMMARY:
the purpose of this study is to determine whether calcium supplementation is effective to prevent preeclampsia in Sichuang Province of china and which dose is more suitable

ELIGIBILITY:
Inclusion Criteria:

* Nulliparity;age ≥35 years;Previous pre-eclampsia;Family history of pre-eclampsia;Multiple pregnancy;Time between pregnancies ≥10years;Body mass index ≥25;diastolic pressure ≥ 80 mm Hg before 20 weeks' gestation;Proteinuria ≥+ on more than one occasion or ≥ 300 mg/24 h before 20 weeks' gestation;Underlying medical conditions(Pre-existing hypertension;Pre-existing renal disease;Pre-existing diabetes;Presence of antiphospholipid antibodies;Chronic autoimmune disease);male sex partner's predecessor wife has Previous pre-eclampsia

Exclusion Criteria:

* first prenatal visit after 16 weeks' gestation;severe anemia;other Underlying medical conditions which need treatment first (such as uncontrolled hyperthyreosis )

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11000 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
incidence of pre-eclampsia | postpartum forty-two days

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu, China